CLINICAL TRIAL: NCT06444620
Title: Efficacy, Safety and Tolerability of Switching to DTG/3TC Single Tablet Regimen From B/F/TAF in Older Persons Living With HIV in Kenya
Brief Title: B/F/TAF to DTG/3TC Switch Study
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University of Nairobi (Other)
Collaborators: ViiV Healthcare (Industry)
Responsible Party: Principal Investigator, Loice Achieng Ombajo, Principal Investigator, University of Nairobi
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Sungura Study
Record Dates: First submitted 2024-05-22; First posted 2024-06-05 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-09

CONDITIONS: HIV-1-infection
Keywords: HIV; Bictegravir; Tenofovir alafenamide; Dolutegravir; Dual therapy; First-line; Elderly; Switch

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Switch to DTG/3TC 2DR (Experimental): Participants will be switched from B/F/TAF to a fixed-dose combined DTG/3TC pill each containing 50mg of dolutegravir and 300mg of lamivudine taken once daily for the duration of the study
  Interventions: Drug: DTG/3TC

INTERVENTIONS:
Drug: DTG/3TC — This is a fixed-dose combined DTG/3TC pill each containing 50mg of dolutegravir and 300mg of lamivudine
  Other Names: Avridela

SUMMARY:
OBJECTIVE:

To assess the efficacy and safety of switch to dolutegravir and lamivudine (DTG/3TC) single tablet regimen from bictegravir, emtricitabine and tenofovir alafenamide (B/F/TAF) in persons living with HIV aged 60 years old or more.

METHODS:

This is a phase 3b, multi-center, open-label, single-arm clinical trial over 96 weeks. The study will take place at two sites in Kenya: Kenyatta National Hospital (KNH) and Jaramogi Oginga Odinga Teaching and Referral Hospital (JOOTRH). Study visits will take place at screening, baseline, and weeks 4, 12, 24, 36, 48, 60, 72, 84, and 96 (with a 6-week extension as required for confirming HIV-1 RNA levels). A target of 240 participants from the ongoing B/F/TAF Elderly Switch Study will be enrolled. Eligible participants will be switched from B/F/TAF to DTG/3TC at enrollment and followed up for 96 weeks. The primary endpoint will be the proportion of participants with plasma HIV-1 RNA ≥ 50 copies/mL (Snapshot algorithm) at Week 48. Analysis of the primary endpoint will be performed for the intention to treat - exposed (ITT-E) population using the FDA snapshot method.

DETAILED DESCRIPTION:
BACKGROUND:

Three drug regimens for the treatment of HIV are widely used and successful in achieving viral suppression. However, they are associated with various adverse events including renal and bone disease, anaemia, mitochondrial toxicity, and possible association with increased cardiovascular events. Data from the ongoing B/F/TAF Elderly Switch Study has demonstrated high rates of renal insufficiency and osteoporosis in people living with HIV aged 60 years or more, hence the need for safe treatment options. Two drug regimens (2DR) have demonstrated non-inferiority to three drug regimens in patients who are treatment-naïve as well as in those who are virally suppressed on a first-line regimen and potentially have lower toxicity, fewer adverse drug events and a lower drug burden.

OVERALL STRATEGY:

This is a phase 3b, multi-centre, open-label, single-arm clinical trial over 96 weeks describing the efficacy of switching virally suppressed HIV-1 infected adults to DTG/3TC dual therapy from their current B/F/TAF regimen. The primary efficacy endpoint is the proportion of participants with viral load (VL) ≥ 50 copies/ml at week 48.

The study will take place at two sites in Kenya: Kenyatta National Hospital (KNH, the largest teaching and referral hospital in Kenya), and Jaramogi Oginga Odinga Teaching and Referral Hospital (JOOTRH, the largest teaching and referral hospital in the Nyanza region of Kenya). The outpatient HIV clinics at these sites currently provide antiretroviral therapy (ART) to over 15,000 persons living with HIV (PWH) combined. These two sites are currently participating in the B/F/TAF-elderly study.

Study visits will take place at screening, baseline, and weeks 4, 12, 24, 36, 48, and 96 (with a 6-week extension as required for confirming HIV-1 RNA levels within the FDA snapshot window). HIV-1 RNA viral load will be performed at screening and weeks 4, 12, 24, 48 and 96. If HIV-1 RNA is ≥ 50 copies/ml then a repeat test will be performed at least 2 weeks after the detectable result to confirm virological failure. If the repeat HIV-1 RNA result is ≥ 50 copies/ml this confirms protocol-defined virological failure (PDVF) and genotypic resistance testing will be performed for any repeat viral load ≥ 500 copies/ml. Other routine study investigations will include CD4 count, complete blood count, serum Cr, renal biomarkers, alanine transaminase (ALT), aspartate aminotransferase (AST), fasting lipids, fasting glucose and patient satisfaction questionnaires (HIVTSQ).

METHODS:

The anticipated sample size is 240 participants started on study treatment among patients on B/F/TAF therapy for at least 24 weeks and no prior virological failure (defined as two consecutive HIV-1 RNA viral loads ≥ 50 copies/ml separated by at least 2 weeks), with a viral load of < 50 copies/ml for at least 12 weeks, and aged 60 years or above.

All participants will be recruited from the pool of patients who are exiting the B/F/TAF-elderly trial at the two study sites. Those who provide written informed consent will be assessed for eligibility through review of their medical records, history and physical examination.

Patients who provide informed consent and meet all eligibility criteria after screening investigations will be enrolled in the study within 28 days of the screening investigations and will complete baseline investigations (CD4 count, fasting lipid profile and fasting glucose). During the enrollment visit participants will be switched to DTG/3TC two drug regimen.

Participants will be engaged in the study for 96 weeks plus up to 28 days between screening and enrolment, and a follow-up visit up to 28 days beyond the week 96 visit if required to confirm HIV-1 RNA within the FDA snapshot window.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to understand and comply with the protocol requirements, instructions and restrictions
* Able and willing to give informed consent
* Have been randomised to the B/F/TAF arm and completed the B/F/TAF-elderly study. Participants should be on B/F/TAF until day 1 of entry into the current study
* HIV-1 RNA viral load < 50 copies/ml at screening (within 28 days prior to enrollment)

Exclusion Criteria:

* Confirmed treatment failure as defined by two consecutive HIV-1 RNA viral loads ≥ 50 copies/ml separated by at least 2 weeks, after at least 6 months on ART or after a documented HIV-1 RNA viral load < 50 copies/ml
* Using any protocol-defined prohibited medicine where the participant is unwilling or unable to switch to an alternative (see Section 5.2. under Prohibited medications and non-drug therapies)
* Evidence of hepatitis B virus (HBV) infection based on the results of testing at screening for hepatitis B surface antigen (HBsAg), hepatitis B core antibody (anti-HBc), hepatitis B surface antibody (anti-HBs) and HBV DNA as follows:

  1. Participants positive for HBsAg are excluded;
  2. Participants negative for anti-HBs but positive for anti-HBc (negative HBsAg status), whether negative or positive for HBV DNA, are excluded;
  3. Participants positive for anti-HBc (negative HBsAg status) and positive for anti-HBs (past and/or current evidence) are immune to HBV and are not excluded.
* Has AST and/or ALT at least 5-times greater than the upper limit of normal
* Severe hepatic impairment (Class C) as determined by Child-Pugh classification
* Has an estimated creatinine clearance (CrCl) below 30 ml/min (as estimated using the Cockcroft-Gault estimate for glomerular filtration rate)
* Documented opportunistic infection within 4 weeks prior to the study enrolment
* Any condition (including illicit drug use or alcohol abuse) or laboratory results which, in the investigator's opinion, interfere with assessments or completion of the study
* Untreated syphilis infection (positive rapid plasma reagin [RPR] at Screening without clear documentation of treatment). Participants who are at least 7 days post completed treatment are eligible.
* History or presence of allergy or intolerance to the study treatment or their components or drugs of their class or a history of drug or other allergy that, in the opinion of the investigator or Medical Monitor, contraindicates their participation.
* Ongoing malignancy other than cutaneous Kaposi's sarcoma, basal cell carcinoma, or resected, non-invasive cutaneous squamous cell carcinoma, or cervical, anal or penile intraepithelial neoplasia.
* Participants who in the investigator's judgment, poses a significant suicidality risk. Participant's history of suicidal behavior and/or suicidal ideation should be considered when evaluating for suicide risk
* Any evidence of any major 3TC resistance associated mutations (M184V/I and/or K65R and/or MDR) or presence of any major INSTI resistance associated mutation

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 240 (Estimated)
Dates: Start 2024-07-22 (Actual); Primary Completion 2025-12-22 (Estimated); Study Completion 2026-12-22 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants with virological failure at week 48 | 48 weeks
  Number and proportion of participants with plasma HIV-1 RNA ≥ 50 copies/mL as per the FDA Snapshot algorithm) at Week 48

SECONDARY OUTCOMES:
Proportion of participants with virological failure at week 24 | 24 weeks
  Number and proportion of participants with plasma HIV-1 RNA ≥ 50 copies/mL as per the FDA Snapshot algorithm at 24 weeks
Proportion of participants with virological failure at week 96 | 96 weeks
  Number and proportion of participants with plasma HIV-1 RNA ≥ 50 copies/mL as per the FDA Snapshot algorithm at 96 weeks
Proportion of participants with treatment success | 24, 48 and 96 weeks
  Number and proportion of participants with plasma HIV-1 RNA <50 copies/mL as per the FDA Snapshot algorithm at 24, 48 and 96 weeks
Change in CD4 | 24, 48 and 96 weeks
  Absolute values and changes from baseline in CD4+ cells count and CD4:CD8 ratio at 24, 48 and 96 weeks
Number of participants with HIV disease progression | 24, 48 and 96 weeks
  Occurrence of disease progression (HIV associated conditions, AIDS, and death) through Weeks 24, 48 and 96
Change in lipid parameters | 24, 48 and 96 weeks
  Change in lipid parameters (total cholesterol, HDL and LDL cholesterol, triglyceride and TC/HDL ratio) from baseline to weeks 24, 48 and 96
Change in fasting blood sugar | 48 and 96 weeks
  Change in fasting blood sugar from baseline to weeks 48 and 96
Change in blood pressure | 24, 48 and 96 weeks
  Change in blood pressure over 24, 48 and 96 weeks
Change in weight | 24, 48 and 96 weeks
  Mean change in weight at week 24, 48 and 96
Change in fat and lean mass | 96 weeks
  Change from baseline in total and regional (trunk and limbs) fat and lean (fat-free) mass by dual energy x-ray absorptiometry (DXA) at 96 weeks in a subset of participants performing DXA scans
Weight gain of 10% or more | 48 and 96 weeks
  Proportion of participants with ≥10% weight gain at weeks 48 and 96
Change in the Atherosclerotic Cardiovascular Disease (ASCVD) score which is a 10-year risk for ASCVD estimation with <5% being low risk and a higher percentage representing increased ASCVD risk | 48 and 96 weeks
  Change from baseline in ASCVD score at weeks 48 and 96
Patient satisfaction as measured using the HIV Treatment Satisfaction Questionnaire - Status version (HIVTSQs) which scores 10 variables on a 7-point likert score ranging from 0 to 6 with a higher score representing a better outcome | 24 and 96 weeks
  Patient satisfaction (HIVTSQs) at baseline, weeks 24 and 96
Change in patient satisfaction as measured using the HIV Treatment Satisfaction Questionnaire - Change version (HIVTSQc) which scores 10 variables on a 7-point likert score ranging from -3 to +3 with a higher score representing a better outcome | 48 weeks
  Patient satisfaction (HIVTSQc) at week 48
Health related quality of life as measured using the World Health Organization Quality of Life brief questionnaire in HIV population (WHOQOL-HIV BREF) tool | 48 and 96 weeks
  Health related quality of life (WHOQOL-HIV BREF) at baseline, week 48 and week 96 assessing 31 aspects on a 5-point likert scale ranging from 1 to 5 with a higher score representing a better outcome
HIV drug resistance | 24, 48 and 96 weeks
  Occurrence of viral resistance in participants meeting confirmed virologic withdrawal criterion (Plasma HIV-1 RNA ≥ 200 copies/mL preceded by a Plasma HIV-1 RNA ≥ 50 copies/mL) over time
Incidence of adverse events | 24, 48 and 96 weeks
  Incidence and severity of adverse events and laboratory abnormalities over time through Week 96
Treatment-related adverse events | 24, 48 and 96 weeks
  Occurrence of DTG/3TC-non-serious adverse drug-related reactions, all serious adverse events and proportion of participants who discontinue treatment due to adverse event
Change in beta-2 microglobulin | 48 and 96 weeks
  Change from Baseline (Day 1) in renal biomarkers at Weeks 48 and 96
Change in retinol binding protein | 48 and 96 weeks
  Change from Baseline (Day 1) in renal biomarkers at Weeks 48 and 96
Change in cystatin C | 48 and 96 weeks
  Change from Baseline (Day 1) in renal biomarkers at Weeks 48 and 96
Change in the estimated glomerular filtration rate as measured using the 2021 CKD-EPI creatinine calculator | 48 and 96 weeks
  Changes from baseline in estimated glomerular filtration rate (CKD-EPI creatinine) at 48 and 96 weeks
Change in the estimated glomerular filtration rate as measured using the 2021 CKD-EPI creatinine-cystatin C calculator | 48 and 96 weeks
  Changes from baseline in estimated glomerular filtration rate (CKD-EPI Creatinine-Cystatin C) at 48 and 96 weeks
Change in urinary protein/creatinine ratio | 48 and 96 weeks
  Changes from baseline in the urinary protein/creatinine at 48 and 96 weeks
Change in AST, ALT and gamma-glutamyltransferase (GGT) | 48 and 96 weeks
  Change from baseline in AST, ALT and GGT levels at week 48 and 96

CONTACTS AND LOCATIONS:
Overall Officials: Loice A Ombajo, MD, MSc, Principal Investigator — University of Nairobi
Locations (2):
- Kenya (2):
  - Jaramogi Oginga Odinga Teaching and Referral Hospital, Kisumu
  - Kenyatta National Hospital, Nairobi

IPD SHARING:
Plan to Share IPD: Yes
We will share the individual patient data (IPD) that underlie the results reported after de-identification (text, tables, figures and appendices)
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: Beginning 6 months after publication of the final manuscript and for a period of 36 months
Access Criteria: Access to IPD will be subject to the University of Nairobi data sharing requirements. Written requests should be submitted to the Principal Investigator providing a brief description of the individual or group making the request and detailing the reason for the same. Prior to sharing the data, the requestor will be required to sign a data access and sharing agreement.